CLINICAL TRIAL: NCT00372489
Title: An Open-Label, Multi-Center, Extension Study to Evaluate the Safety and Tolerability of Peginesatide for the Long-Term Maintenance Treatment of Anemia in Patients With Chronic Kidney Disease
Brief Title: Extension Study to Evaluate Safety and Tolerability of Peginesatide for Long-Term Treatment of Anemia in Participants With CKD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to more robust long-term data generated in other active-controlled studies
Sponsor: Affymax (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-09
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Results first posted 2012-05-28 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemodialysis; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — peginesatide; hematide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peginesatide (Experimental)
  Interventions: Drug: peginesatide

INTERVENTIONS:
Drug: peginesatide — Participants received the same initial peginesatide dose as was administered at the end of the previous peginesatide treatment study (NCT00228449) in which the participant was enrolled. The median first dose at study start was 0.087 milligram per kilogram (mg/kg) with an interquartile range of 0.064 to 0.123 mg/kg. Each participant was to receive peginesatide as an injection administered intravenously once every 4 weeks for approximately 54 months in this trial.
  Other Names: Omontys; Hematide; AF37702 Injection

SUMMARY:
The purpose of this study was to evaluate the long term safety and tolerability of peginesatide for the maintenance of hemoglobin in participants with chronic kidney disease (CKD) who had received at least 24 weeks of peginesatide treatment in an earlier study.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents have been established as a treatment for anemia in subjects with chronic kidney disease, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia associated with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor, and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents (ESAs).

Study participants had received at least 24 weeks of peginesatide dosing in a previous Affymax-sponsored study (NCT00228449) and were to receive doses of peginesatide for approximately 54 months. However, the Sponsor ended the study early.

ELIGIBILITY:
Inclusion Criteria:

* Participant is informed of the investigational nature of this study and has given written, witnessed informed consent in accordance with institutional, local, and national guidelines
* Males or females ≥ 18 years of age. Pre-menopausal females (with the exception of those who are surgically sterile) must have a negative pregnancy test at screening; those who are sexually active must practice a highly effective method of birth control for at least 4 weeks prior to study drug administration, and must be willing to continue contraception until at least 4 weeks after the last dose of study drug.
* Participant who has received at least 24 weeks of peginesatide dosing in a previous Affymax-sponsored study
* One hemoglobin value of > 10.0 g/dL in the 4 weeks prior to study drug administration

Exclusion Criteria:

* Known intolerance to peginesatide or pegylated products
* History of antibodies to any erythropoiesis stimulating agent (ESA) or history of pure red cell aplasia (PRCA)
* High likelihood of early withdrawal or interruption of the study (e.g., participant suffers from any clinically significant medical disease or condition that may, in the Investigator's opinion, interfere with safety, assessment, or follow-up of the participant)
* Anticipated life expectancy < 18 months
* Receipt of any ESA other than peginesatide at any time after participant enrollment in the previous Affymax-sponsored study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (9):
- United States (9):
  - Research Facility, Pine Bluff, Arkansas
  - Research Facility, Mountain View, California
  - Research Facility, Lauderdale Lakes, Florida
  - Research Facility, Pembroke Pines, Florida
  - Research Facility, Shreveport, Louisiana
  - Research Facility, Detroit, Michigan
  - Research Facility, Canton, Ohio
  - Research Facility, Nashville, Tennessee
  - Research Facility, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peginesatide
Started | 81
Completed | 2
Not Completed | 79
Not completed — Adverse Event | 18
Not completed — Lack of Efficacy | 1
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 5
Not completed — Patient Relocation | 2
Not completed — Renal transplant | 6
Not completed — Sponsor Decision to Terminate Study | 41

BASELINE CHARACTERISTICS:
Arm/Group | Peginesatide
Number analyzed (Participants) | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 59.8 (15.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 44

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Mean Hemoglobin in the Target Range of 10.0-12.0 Grams Per Deciliter (g/dL) After Dosing Guideline Change
Time Frame: Up to 54 months
Population: Full Analysis - Number of participants with hemoglobin assessed after dosing guideline change
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide
Number analyzed (Participants) | 60
percentage of participants | 0.867

ADVERSE EVENTS:
Arm/Group | Peginesatide
Serious Adverse Events (participants affected / at risk) | 58/81
Other Adverse Events (participants affected / at risk) | 77/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=81)
Anaemia (Blood and lymphatic system disorders) | 6
Cardiac failure congestive (Cardiac disorders) | 16
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4
Chest pain (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Sarcoidosis (Immune system disorders) | 1
Pneumonia (Infections and infestations) | 9
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3
Fluid overload (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Syncope (Nervous system disorders) | 3
Mental status changes (Psychiatric disorders) | 2
Renal failure chronic (Renal and urinary disorders) | 3
Balanitis (Reproductive system and breast disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Swelling face (Skin and subcutaneous tissue disorders) | 1
Hypertensive crisis (Vascular disorders) | 4
Acute myocardial infarction (Cardiac disorders) | 9
Gastritis (Gastrointestinal disorders) | 2
Non-cardiac chest pain (General disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Sepsis (Infections and infestations) | 5
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 4
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 3
Coronary artery disease (Cardiac disorders) | 5
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2
Catheter related complication (General disorders) | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Gangrene (Infections and infestations) | 4
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Dementia (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 3
Atrial fibrillation (Cardiac disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Arteriovenous graft site infection (Infections and infestations) | 3
Acetabulum fracture (Injury, poisoning and procedural complications) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Dizziness (Nervous system disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Deep vein thrombosis (Vascular disorders) | 2
Myocardial infarction (Cardiac disorders) | 4
Ascites (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Bacteraemia (Infections and infestations) | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Lactose intolerance (Metabolism and nutrition disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 2
Cardio-respiratory arrest (Cardiac disorders) | 3
Colitis (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 3
Arteriovenous graft aneurysm (Injury, poisoning and procedural complications) | 1
Migraine (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Aortic dissection (Vascular disorders) | 1
Angina pectoris (Cardiac disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 1
Polyneuropathy (Nervous system disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Bradycardia (Cardiac disorders) | 2
Gastric ulcer (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
Presyncope (Nervous system disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 2
Gastritis erosive (Gastrointestinal disorders) | 1
Clostridium difficile colitis (Infections and infestations) | 2
Hip fracture (Injury, poisoning and procedural complications) | 1
Transient ischaemic attack (Nervous system disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Bronchitis (Infections and infestations) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Lymphocele (Vascular disorders) | 1
Angina unstable (Cardiac disorders) | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1
Catheter sepsis (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Atrial thrombosis (Cardiac disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Escherichia sepsis (Infections and infestations) | 1
Sternal injury (Injury, poisoning and procedural complications) | 1
Cardiac arrest (Cardiac disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Extradural abscess (Infections and infestations) | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1
Cardiogenic shock (Cardiac disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Graft infection (Infections and infestations) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Cardiomyopathy (Cardiac disorders) | 1
Lobar pneumonia (Infections and infestations) | 1
Pericardial effusion (Cardiac disorders) | 1
Postoperative wound infection (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 1
Pyelonephritis (Infections and infestations) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Septic shock (Infections and infestations) | 1
Ventricular arrhythmia (Cardiac disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Ventricular fibrillation (Cardiac disorders) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Streptococcal sepsis (Infections and infestations) | 1
Tubo-ovarian abscess (Infections and infestations) | 1
Urosepsis (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=81)
Anaemia (Blood and lymphatic system disorders) | 10
Tachycardia (Cardiac disorders) | 7
Hyperparathyroidism (Endocrine disorders) | 6
Conjunctivitis (Eye disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 20
Vomiting (Gastrointestinal disorders) | 16
Nausea (Gastrointestinal disorders) | 13
Dyspepsia (Gastrointestinal disorders) | 9
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 5
Pyrexia (General disorders) | 16
Oedema peripheral (General disorders) | 12
Chest pain (General disorders) | 11
Asthenia (General disorders) | 8
Chest discomfort (General disorders) | 8
Fatigue (General disorders) | 7
Chills (General disorders) | 6
Pain (General disorders) | 5
Upper respiratory tract infection (Infections and infestations) | 23
Nasopharyngitis (Infections and infestations) | 14
Sinusitis (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 23
Vascular graft complication (Injury, poisoning and procedural complications) | 15
Procedural hypotension (Injury, poisoning and procedural complications) | 12
Fall (Injury, poisoning and procedural complications) | 6
Procedural headache (Injury, poisoning and procedural complications) | 6
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 5
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 5
Procedural dizziness (Injury, poisoning and procedural complications) | 5
Wound (Injury, poisoning and procedural complications) | 5
Breath sounds abnormal (Investigations) | 7
Hyperphosphataemia (Metabolism and nutrition disorders) | 14
Iron deficiency (Metabolism and nutrition disorders) | 13
Hyperkalaemia (Metabolism and nutrition disorders) | 11
Hypercalcaemia (Metabolism and nutrition disorders) | 9
Hyperlipidaemia (Metabolism and nutrition disorders) | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 6
Muscle spasms (Musculoskeletal and connective tissue disorders) | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 10
Dizziness (Nervous system disorders) | 10
Headache (Nervous system disorders) | 10
Hypoaesthesia (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 11
Anxiety (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20
Cough (Respiratory, thoracic and mediastinal disorders) | 12
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9
Hypertension (Vascular disorders) | 10
Hypotension (Vascular disorders) | 6

LIMITATIONS AND CAVEATS:
Early termination of study due to generation of controlled long-term data in Phase 3 studies. Amended dosing guidelines during the trial to reflect label changes for ESAs; the primary outcome was assessed after the dosing guideline change.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications may not contain Sponsor confidential information, and may be subject to Sponsor review 30 days prior to submission for publication.